CLINICAL TRIAL: NCT00050947
Title: A Multicenter, Rater-blind, Randomized, Age-stratified, Parallel-group Study Comparing Two Doses of Oxcarbazepine as Monotherapy in Pediatric Patients With Inadequately-controlled Partial Seizures.
Brief Title: Pediatric Epilepsy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Purpose: Treatment
Other Study IDs: CTRI476E2339
Record Dates: First submitted 2002-12-30; First posted 2003-01-01 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Epilepsy
Keywords: partial seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Oxcarbazepine

INTERVENTIONS:
Drug: oxcarbazepine

SUMMARY:
This study will evaluate the safety and effectiveness of oxcarbazepine (Trileptal) as monotherapy in the treatment of partial seizures in pediatric patients 1 month to 3 years of age.

ELIGIBILITY:
INCLUSION CRITERIA: To enter this study, patients must:

* Have a diagnosis of partial seizures
* Have 2-30 seizures per week while on a stable dose of one anti-epileptic drug or be a patient recently diagnosed with partial seizures and currently receiving no seizure medication
* Be willing to be hospitalized for up to 5 days
* Weigh a minimum of 6.6 lbs
* Have had a previous CAT scan/MRI confirming the absence of space occupying lesions or progressive neurological disease
* Have normal laboratory results

EXCLUSION CRITERIA: To enter this study, a patient must not have or be:

* Seizures caused by metabolic disturbance, toxic exposure, or active infection
* A primary diagnosis of generalized epilepsy (exception - secondarily generalized seizures)
* A history of status epilepticus within 30 days
* Seizures not related to epilepsy
* This study has some AED restrictions
* Serum sodium levels <135 mEq/L
* Significant heart, breathing, kidney, stomach, liver, blood, or cancer disorder requiring treatment/therapy
* A history of chronic infection (e.g., hepatitis or HIV)
* Significant electrocardiogram (ECG) abnormalities
* A nursing mother taking anti-convulsant drugs
* A history of substance abuse (including alcohol)
* Previously demonstrated sensitivity/allergic reaction to Trileptal or related compounds
* Used experimental medication within 30 days of entering this study

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2002-07; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Time to meeting one of the exit criteria starting from the first dose of oxcarbazepine on Day 3.

SECONDARY OUTCOMES:
Percentage of patients meeting one of the exit criteria and the electrographic partial seizure frequency/24 hours during the treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (25):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Madera, California
  - Orange, California
  - Denver, Colorado
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Ann Arbor, Michigan
  - Duluth, Minnesota
  - Saint Paul, Minnesota
  - Chesterfields, Missouri
  - St Louis, Missouri
  - Buffalo, New York
  - New York, New York
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Spartenberg, South Carolina
  - Fort Worth, Texas
  - Houston, Texas
- Brigadeiro Hospital, Sao Paulo - SP, Brazil
- Germany (3):
  - Jena
  - Kehl-Kork
  - Kiel
- Novartis, Mexico City, Mexico